CLINICAL TRIAL: NCT01468571
Title: Effects of Spironolactone on Collagen Metabolism in Pulmonary Arterial Hypertension
Brief Title: Effects of Spironolactone on Collagen Metabolism in Patients With Pulmonary Arterial Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Zeenat Safdar, Associate Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H24178; K23HL093214 (NIH)
Record Dates: First submitted 2011-11-03; First posted 2011-11-09 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Pulmonary Hypertension
Keywords: Potassium Sparing Diuretics; Right-sided heart failure; Edema
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure; Edema | interventions — Spironolactone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Experimental): Drug: Spironolactone Drug: Placebo
  Interventions: Drug: Spironolactone
- Placebo (Experimental): Drug: Placebo Drug: Spironolactone
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 50 mg po daily of spironolactone for 8 weeks. A cross-over study where each subject will receive spironolactone or placebo in a random order for 8 weeks each.
  Other Names: Aldactone
  Arms: Spironolactone
Drug: Placebo — Each subject will receive placebo or spironolactone for 8 weeks. At the end of week 8, treatment arm for each subject will be blindly switched.
  So if a study patient received placebo for the first 8 weeks then he/she will be switched to receive active drug (spironolactone) for the next 8 weeks.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of spironolactone on collagen markers in a large number of patients with pulmonary hypertension. In addition, safety and tolerability of spironolactone, an aldosterone receptor antagonist, in patients with pulmonary arterial hypertension, will be determined.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is an orphan disease characterized by pulmonary artery hypertrophy, and resulting vascular remodeling of involved vessels, often leading to right heart failure. Accumulating evidence from vascular biology, animal models, and therapeutic drug trials suggests significant contributions of the neurohormonal milieu to the disease process, morbidity, and mortality. The renin-angiotensin-aldosterone system (RAAS) is an important neurohormonal pathway that induces collagen synthesis in the myocardium and systemic vasculature. There is paucity of data regarding the contribution of RAAS in the pathogenesis of PAH and the effects of aldosterone blockade in the amelioration of PAH. Thus, the overall goal of this proposal is to investigate the contribution of RAAS to the pathogenesis of PAH, and to explore the effects of an aldosterone blocker, spironolactone, in PAH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Body weight > 40 kg
* PAH Diagnostic Group I
* Stable subjects with no change in PAH specific therapy within the last 4 weeks
* No change in dose of background therapy (digoxin, diuretic) within the last 2 weeks excluding anticoagulation

Exclusion Criteria:

* Unable to give informed consent
* Hemodynamically unstable subjects
* Pregnant or breast feeding
* Have significant renal insufficiency (serum creatinine >2.5 mg per deciliter or required hemodialysis)
* Have significant liver dysfunction (AST or ALT more than three times upper limit of normal)
* Currently on aldosterone receptor blocker (spironolactone or eplerenone) or ACE inhibitor
* PH due to left heart disease
* Unable or unwilling to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in biomarker levels in the spironolactone treated as compared to placebo treated group. | 16 week
  50 participants will be enrolled in a 16-week study, and each subject will receive placebo or active drug in a random order. At the end of week 8, treatment arm for each subject will be blindly switched. Biomarker levels will be drawn 3 times (baseline, week 8, and week 16) during the study period for each subject.

SECONDARY OUTCOMES:
Number of adverse events in patients treated with spironolactone as compared to placebo. | 16 week
  Safety and tolerability of spironolactone as compared to placebo in PAH.
Change in six-minute walk distance from baseline to week 8 and week 16. | 16 week
Composite end-point | 16 week
  Composite end-point predefined as greater than 10% increase in walk distance, improvement by at least one functional class and absence of clinical worsening. Clinical worsening will be defined as hospitalization for worsening PAH, all-cause death, addition of prostacyclin therapy, lung transplantation, or atrial septostomy.

CONTACTS AND LOCATIONS:
Overall Officials: Zeenat Safdar, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States